CLINICAL TRIAL: NCT03856424
Title: Effect of Three Modalities of Spontaneous Breathing Tests on Respiratory Efforts in Tracheostomized Patients. Monocentric Crossover Interventionnal Study.
Brief Title: Effect of Three Modalities of Spontaneous Breathing Tests on Respiratory Efforts in Tracheostomized Patients
Acronym: TWEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Piquilloud Imboden Lise (Other)
Responsible Party: Sponsor-Investigator, Piquilloud Imboden Lise, Sponsor-investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TWEEP
Record Dates: First submitted 2019-01-28; First posted 2019-02-27 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Mechanical Ventilation Complication
Keywords: Ventilation; Tracheotomy; Difficult weaning; Spontaneous Breathing Test; Esophageal pressure; Work of breathing; Esophageal pressure time-product; Difficult weaning from mechanical ventilation; Ventilation weaning
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Three different spontaneous breathing trials modalities will be tested in each patient in a randomized order. Washout periods will be performed between the tested modalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Modality 1 - Washout - Modality 2 - Washout - Modality 3 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3
- Modality 1 - Washout - Modality 3 - Washout - Modality 2 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3
- Modality 2 - Washout - Modality 1 - Washout - Modality 3 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3
- Modality 2 - Washout - Modality 3 - Washout - Modality 1 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3
- Modality 3 - Washout - Modality 2 - Washout - Modality 1 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3
- Modality 3 - Washout - Modality 1 - Washout - Modality 2 (Other): Three different 30-minute modalities of deventilation will be performed in a randomized order in each patient. Washout periods of 30 minutes will occur between tested modalities.
  Interventions: Procedure: Modality 1; Procedure: Modality 2; Procedure: Modality 3

INTERVENTIONS:
Procedure: Modality 1 — Pressure support ventilation (PSV) modality
Procedure: Modality 2 — T-Piece modality
Procedure: Modality 3 — High-flow oxygen

SUMMARY:
Datas are lacking concerning weaning from mechanical ventilation for tracheostomized patients. In particular, the effect of different modalities of spontaneous breathing trials on respiratory effort has not been extensively described.

This crossover physiology study will include 18 tracheostomized patients ventilated for more than 72 hours.

The objective of this study is to compare the effect of three different modalities of SBTs on respiratory effort in tracheostomized patients. The modalities tested are : Pressure Support Ventilation (PSV level 5 cmH2O, PEEP 5 cmH2O), T-piece test and high-flow Oxygen. Each modality is applied in a randomized order, during 30 minutes. During every modality tested, esophageal and gastric pressure, expired CO2, and comfort will be monitored, in addition to standard monitoring. Based on esophageal pressure monitoring, patient's respiratory efforts can be calculated either by esophageal pressure-time product and work of breathing. Pressure generated by inspiratory muscles will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a tracheostomy is planned
* Patients on invasive ventilation for >72 hours

Exclusion Criteria:

* Tracheostomy for upper airway obstruction or other disease
* Patients tracheostomized before current hospitalization
* Patients with Glasgow Coma Scale (GCS) < 8/10 after cardiac arrest
* Patients with GCS < 8/10 because of primary central neurologic disease
* Patients for whom therapeutic limitations have already been decided
* Patients for whom weaning from ventilation is not an objective
* Patients suffering from myasthenia gravis
* Patients with cardiac assistance device
* Patients with medullary lesion proximal to C5
* Patients for whom nasogastric tube insertion is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of pressure-time product of esophageal pressure | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Quantification of inspiratory effort of the patient

SECONDARY OUTCOMES:
Evolution of work of breathing (WOB) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Total area of a Campbell diagram for esophageal pressure and volume during one respiratory cycle
Evolution of esophageal pressure drop | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Maximum variation of esophageal pressure during respiratory cycles
Evolution of inspiratory muscle pressure (Pmus) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Pressure generated by patients' respiratory muscles
Evolution of transdiaphragmatic pressure (Ptransdiaph) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Difference between gastric and esophageal pressure. Reflect of pressure generated by diaphragm during inspiration
Evolution of tidal volume (VT) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
Evolution of respiratory rate (RR) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
Evolution of inspiratory airway flow | Recorded every 5 minutes during each sequence and washout period, 180 minutes
Evolution of ratio of inspiratory time over total duration of a breathing cycle (ti/ttot) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
Evolution of Rapid Shallow Breathing Index (RSBI) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  RR/VT - predictor during ventilation weaning of intolerance of SBT
Evolution of respiratory system compliance (Crs) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Capacity of total respiratory system to gain volume for a given pressure
Evolution of lungs compliance (CL) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Capacity of lungs to gain volume for a given pressure
Evolution of chest wall compliance (Ccw) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Capacity of lungs to gain volume for a given pressure
Evolution of transpulmonary pressure (Ptranspulm) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Alveolar pressure minus pleural pressure
Evolution of ratio of total dead space volume over tidal volume | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Calculated by means of expired CO2 and arterial blood gas CO2
Evolution of total dead space volume | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Calculated by means of expired CO2
Evolution of total Positive End-Expiratory Pressure (PEEPtot) | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Airway pressure during end-expiratory ventilator occlusion
Evolution of heart rate | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Standard monitoring
Evolution of blood pressure | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Standard monitoring
Evolution of Plateau pressure (Pplat) | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Airway pressure during end-inspiratory ventilator occlusion (corresponds to alveolar pressure)
Evolution of intrinsic Positive End-Expiratory Pressure (PEEPi) | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  PEEPi minus PEEP set on ventilator
Pulmonary strain | Recorded every 5 minutes during each sequence and washout period, 180 minutes
  Measured as the ratio of tidal volume over functionnal residual capacity (FRV)
Evolution of Diaphragmatic excursion (DE) | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Ultrasound measurement of diaphragm movement during inspiration
Evolution of Diaphragmatic thickening fraction (DTF) | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Ultrasound measurement of diaphragm thickening during inspiration
Evolution of hematocrits | Recorded at minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Mesured by arterial blood
Evolution of Richmond Agitation/Sedation scale (RASS) score | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Used in ICU to monitor neurologic changes in patients. Scale from -5 (unarousable) to +4 (combative). 0 is a calm and responsive patient.
Evolution of Borg dyspnea scale score | Recorded at minute 1 and minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Numeric scale to quantify dyspnea from 0 to 10. 0 mean patient does not feel that breathing is difficult and 10 is a maximal dyspnea.
  Measured twice during each Spontaneous Breathing Trial
Evolution of Multidimensionnal dyspnea scale (MDP) score | Recorded at minute 30 of each three spontaneous Breathing Trial, 90 minutes
  Score to quantify comfort, dyspnea and assess respiratory effort as perceived by patient. This scale contains multiple items, divided in two dimensions : sensory and affective.
  Sensory dimension contains : intensity on a scale of 0 to 10 of five sensory qualities (physical breathing effort, air hunger, tightness, mental breathing effort, hyperpnoea) Affective dimension contains : a breathing discomfort scale (scale of 0 to 10)
  Measured once during each Spontaneous Breathing Trial

CONTACTS AND LOCATIONS:
Overall Officials: Lise Piquilloud Imboden, MER&PD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided